CLINICAL TRIAL: NCT00376051
Title: Serotonergic Function and Behavioural and Psychological Symptoms of Frontotemporal Dementia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Alzheimer Society of Canada (Other)
Responsible Party: Dr. Nathan Herrmann, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 218-2006; 07-48
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2009-11

CONDITIONS: Frontotemporal Dementia
Keywords: frontotemporal lobar degeneration; frontotemporal dementia; serotonin; dementia; behavioural disturbances
MeSH Terms: conditions — Frontotemporal Dementia; Frontotemporal Lobar Degeneration; Dementia; Mental Disorders | interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Citalopram — Titrates from 10mg/day to 40mg/day, increases 10mg per week.

SUMMARY:
Frontotemporal lobar degeneration(FTLD) is a common cause of early-onset dementia. FTLD is characterized multiple behavioral symptoms including mental rigidity, irritability, emotional blunting, disinhibition, apathy, and aggression. These behavioural disturbances are particularly important because they increase caregiver burden and may lead to earlier institutionalization. While the causes of FTLD are largely unknown, there is a great deal of evidence suggesting that a brain chemical called serotonin regulates many of the behaviours that are disturbed in FTLD. Our objective is therefore to determine whether dysfunction in the brain's serotonin system is responsible for behavioural problems among FTLD patients. We hope to take the first steps towards a scientific understanding of the behavioural symptoms of FTD, and use our findings to support a larger study optimizing the treatment of targeted behavioural disturbances in FTLD using the antidepressant citalopram.

Citalopram increases transmission by serotonin; we plan to use this medication to determine whether there are any differences in how the serotonin system functions in FTLD patients who display different levels of behavioural disturbances. Patients will be given citalopram and will have their blood drawn after 2 and 3 hours to determine plasma levels of the hormones cortisol and prolactin at those times. These hormones are good indicators of serotonergic functioning in the central nervous system.

We expect that patients with lower levels of serotonergic functioning will have more severe behavioural disturbances and be less responsive to treatment with citalopram. Following their first test day, we will provide patients with a 6-week supply of citalopram, and assess them for any changes in behaviour at the end of this treatment.

This study aims to obtain a better understanding of how changes in the serotonin system relate to behavioural symptoms in FTLD patients. Using the information from this pilot study, we can plan a larger study to determine whether certain behaviours will respond to treatment with citalopram, and if so, determine whether it is possible to predict which patients, based on individual characteristics, are most likely to respond to this treatment. This methodology will therefore not only provide a scientific rationale for treatment of FTLD, but also provide guidance for ongoing, individualized therapy.

DETAILED DESCRIPTION:
Objectives: A hallmark of frontotemporal lobar degeneration(FTLD) is its associated behavioural disturbances (BPSD), which include disinhibition, aggression, apathy, agitation, depression, and inappropriate affect. Current evidence suggests that secondary changes in the serotonergic system may be key to many of the symptoms of FTLD. Our primary objective is to evaluate the ability of serotonergic dysfunction, as measured through oral citalopram challenge, to predict subsequent behavioural response to pharmacotherapy with citalopram. As a secondary objective, we will explore the relationship between specific BPSDs and the level of serotonergic dysfunction.

Hypotheses: We predict that patients with FTLD who respond to citalopram pharmacotherapy will show greater dysfunction in the serotonergic system, as measured by citalopram challenge, than patients who do not respond. This hypothesis will be evaluated in vivo using peak change in plasma concentrations of cortisol and prolactin as indicators of serotonergic dysfunction following oral citalopram challenge.

Research Plan: A consecutive sample of patients attending FTLD clinics who exhibit significant BPSD will be recruited into this study.Because serotonin promotes cortisol and prolactin secretion via the hypothalamic-pituitary-adrenal (HPA) axis, these hormones have been shown to be a reliable marker of serotonergic functioning. Their levels will therefore be measured from blood samples taken at baseline and 2 and 3 hours after the administration of 20 mg citalopram. Changes in cortisol levels after citalopram administration will be used as the primary measure of serotonergic functioning. We expect to find an inverse correlation between the cortisol response to citalopram challenge and the severity of BPSD according to the total Neuropsychiatric Inventory (NPI) score. Subsequent to the citalopram challenge, participants will be treated for their BPSD with open-label citalopram (20-40 mg) for 6 weeks. At the end of this period, patients will be re-assessed with the NPI. The magnitude of response, based on changes in NPI scores, will be correlated with the citalopram challenge test results. It is expected that patients who show more severe serotonergic dysfunction will have a better response to daily citalopram treatment.

Relevance: The results of this study will further the scientific understanding of the neurochemical basis underlying BPSD in FTLD. To date, the treatment of FTLD patients has relied largely on the understanding of treatments for other dementias, due to the lack of research in the area of FTLD. Therefore, our work may aid in the development of targeted therapies specific to FTLD.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-IV criteria for primary degenerative dementia
* Meet standard clinical criteria for frontotemporal dementia (ie., frontotemporal degeneration including both the frontal/behavioural variant and primary progressive aphasia)
* Have significant behavioural problems as demonstrated by a score of at least eight on the Neuropsychiatric Inventory (NPI) an
* An independent clinical decision to receive psychotropic medication for behavioural disorders

Exclusion Criteria:

* An abnormal biochemical screening (blood cell count, vitamin B12 or thyroid function tests)
* Significant medical illness or other medical/neurological conditions which diminish cognitive function (including: drug overdose, severely disturbed liver, kidney, lung or heart function, anemia, hypothyroidism, vitamin B12 or folic acid deficiency, syphilis, uncontrolled diabetes, Parkinson's disease, Huntington's chorea, progressive supranuclear paralysis, brain tumour, subdural hematoma, multiple sclerosis, or brain trauma);
* An Hachinski ischemic score ≥444;
* Electrocardiographic, laboratory or physical evidence of significant cardiovascular disease;
* Hypertension >160 mmHg systolic or >100 mmHg diastolic;
* A brain computed tomographic scan that could not be interpreted as consistent with FTLD;
* Presence of premorbid or current psychiatric diagnosis (including: major depression, schizophrenia, psychotic symptoms of a severity likely to provoke violent or dangerous behaviour such as command hallucinations to harm people or persecutory delusions that provoke violent reactions, psychoactive substance abuse or dependence);
* Contraindications to receiving citalopram (such as concomitant MAOI or within 2 weeks, or hypersensitivity to citalopram); or
* Ongoing need for psychotropic medications (i.e., unsuitable for washout) or administration of a depot antipsychotic injection within one treatment cycle of visit 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory (NPI) | Screening, Baseline, 4 weeks and 6 weeks

SECONDARY OUTCOMES:
Frontal Behavioural Inventory (FBI) | Baseline, 4 weeks, 6 weeks
Clinical Global Impression (CGI) | Screening, 4 week, 6 week
Cornell Scale for Depression in Dementia | Baseline, 4 weeks and 6 weeks
Disability Assessment for Dementia Scale (DAD) | Baseline, 4 weeks and 6 weeks
Functional Assessment Staging (FAST) | Baseline, 4 weeks and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Krista Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre; Nathan Herrmann, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Baycrest Centre for Geriatric Care, Toronto, Ontario

REFERENCES:
- [Result] Herrmann N, Black SE, Chow T, Cappell J, Tang-Wai DF, Lanctot KL. Serotonergic function and treatment of behavioral and psychological symptoms of frontotemporal dementia. Am J Geriatr Psychiatry. 2012 Sep;20(9):789-97. doi: 10.1097/JGP.0b013e31823033f3. PMID 21878805